CLINICAL TRIAL: NCT00404235
Title: A Phase II Trial of Carboplatin (CBDCA) and ABI-007(ABX) in Patients With Unresectable Stage IV Melanoma
Brief Title: Carboplatin and ABI-007 in Treating Patients With Stage IV Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N057E; NCI-2012-02705 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000514561 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Carboplatin; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- paclitaxel + carboplatin (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation (ABI-007) IV over 30 minutes followed by carboplatin IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for at least 8 courses in the absence of disease progression or unacceptable toxicity.
  Blood and tumor tissue samples are collected periodically to evaluate secreted protein acidic and rich in cysteine (SPARC) content of tumor tissue by immunohistochemistry and to explore the impact of therapy on immune homeostasis. Samples are also analyzed by immunoenzyme techniques for angiogenesis markers.
  After completion of study treatment, patients are followed periodically for up to 2 years.
  Interventions: Drug: carboplatin; Drug: paclitaxel albumin-stabilized nanoparticle formulation

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel albumin-stabilized nanoparticle formulation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and ABI-007, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving carboplatin together with ABI-007 works in treating patients with stage IV melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety and antitumor activity of carboplatin and paclitaxel albumin-stabilized nanoparticle formulation (ABI-007) in patients with unresectable stage IV melanoma who have not received prior chemotherapy for their metastatic disease. (Cohort 1)
* Assess the safety and antitumor activity of this regimen in patients with unresectable stage IV melanoma who have received prior chemotherapy for their metastatic disease. (Cohort 2)

Secondary

* Describe the impact of this regimen on parameters of immune function and angiogenesis in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy for metastatic disease (yes vs no).

Patients receive paclitaxel albumin-stabilized nanoparticle formulation (ABI-007) IV over 30 minutes followed by carboplatin IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for at least 8 courses in the absence of disease progression or unacceptable toxicity.

Blood and tumor tissue samples are collected periodically to evaluate secreted protein acidic and rich in cysteine (SPARC) content of tumor tissue by immunohistochemistry and to explore the impact of therapy on immune homeostasis. Samples are also analyzed by immunoenzyme techniques for angiogenesis markers.

After completion of study treatment, patients are followed periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 74 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable stage IV melanoma
* Measurable disease
* Must have formalin-fixed, paraffin-embedded tumor tissue available for secreted protein acidic and rich in cysteine (SPARC) analysis pre-treatment (Mayo Clinic patients must be willing to submit a repeat biopsy at time of tumor progression)
* Brain metastases allowed provided they were previously treated with no progression for ≥ 3 months

  * Patients with known brain metastases may receive concurrent steroid treatment

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (may be transfused to meet this requirement)
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN (elevated bilirubin allowed in patients with documented Gilbert's syndrome)
* AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after completion of study therapy
* No uncontrolled intercurrent illness including, but not limited to, the following:

  * Active infection
  * Congestive heart failure (New York Heart Association class III-IV heart disease)
* No peripheral neuropathy ≥ grade 2
* No other malignancy within the past 5 years except basal cell or squamous cell carcinoma of the skin previously treated with local resection only or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 4 weeks since prior radiotherapy
* At least 4 weeks since prior interferon or interleukin-2
* At least 4 weeks since prior chemotherapy (cohort 1 )
* No prior chemotherapy in the metastatic setting (cohort 2)
* No prior treatment for melanoma with any of the following agents:

  * Platinum chemotherapy (e.g., carboplatin or cisplatin)
  * Taxanes (e.g., paclitaxel or docetaxel)
  * Paclitaxel albumin-stabilized nanoparticle formulation (ABI-007)
* No other concurrent chemotherapy
* No other concurrent investigational agents
* No concurrent radiotherapy, including palliative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic
Locations (156):
- United States (156):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Kottschade LA, Suman VJ, Amatruda T 3rd, McWilliams RR, Mattar BI, Nikcevich DA, Behrens R, Fitch TR, Jaslowski AJ, Markovic SN. A phase II trial of nab-paclitaxel (ABI-007) and carboplatin in patients with unresectable stage IV melanoma : a North Central Cancer Treatment Group Study, N057E(1). Cancer. 2011 Apr 15;117(8):1704-10. doi: 10.1002/cncr.25659. Epub 2010 Nov 8. PMID 21472717

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Prior Chemotherapy, PT): Patients with malignant melanoma who have received prior chemotherapy for their metastatic disease receive 100 mg/m^2 paclitaxel albumin-stabilized nanoparticle formulation (ABI-007) IV over 30 minutes followed by AUC 2 carboplatin IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for at least 8 courses in the absence of disease progression or unacceptable toxicity.
- Cohort 2 (Chemotherapy Naive, CN): For patients with malignant melanoma who have not received prior chemotherapy for their metastatic disease, patients receive 100 mg/m^2 paclitaxel albumin-stabilized nanoparticle formulation (ABI-007) IV over 30 minutes followed by AUC 2 carboplatin IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for at least 8 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort 1 (Prior Chemotherapy, PT) | Cohort 2 (Chemotherapy Naive, CN)
Started | 35 | 41
Completed | 34 | 39
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Prior Chemotherapy, PT) | Cohort 2 (Chemotherapy Naive, CN) | Total
Number analyzed (Participants) | 34 | 39 | 73
Age, Continuous [Median (Full Range); unit: years] | 60 [28 to 84] | 59 [23 to 91] | 59 [23 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 23 | 23 | 46
Region of Enrollment [Number; unit: participants]
  United States | 34 | 39 | 73

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate, as Measured by RECIST Criteria
Description: The RECIST criteria will be used for response assessments. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. A confirmed tumor response is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart. The tumor response rate is defined as the total number of eligible patients who achieved a complete or partial response according to the RECIST criteria divided by the total number of eligible patients enrolled on study. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response.
Time Frame: Up to 2 years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (Prior Chemotherapy, PT) | Cohort 2 (Chemotherapy Naive, CN)
Number analyzed (Participants) | 34 | 39
percentage of participants | 8.8 [2.5 to 21.3] | 25.6 [14.6 to 39.6]

2. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 (Prior Chemotherapy, PT) | Cohort 2 (Chemotherapy Naive, CN)
Number analyzed (Participants) | 34 | 39
months | 10.9 [4 to NA] — At the time follow-up was terminated for this clinical trial, several patients had not yet died. Their survival time will remain unknown and not collected. | 11.1 [1 to NA] — At the time follow-up was terminated for this clinical trial, several patients had not yet died. Their survival time will remain unknown and not collected.

3. Secondary Outcome: Time to Disease Progression
Description: Time-to-disease progression (TTP) is defined as the time from registration to documentation of disease progression. If a patient dies without a documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death. The distribution of time-to-progression will be estimated using the method of Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 (Prior Chemotherapy, PT) | Cohort 2 (Chemotherapy Naive, CN)
Number analyzed (Participants) | 34 | 39
months | 4.1 [1 to NA] — At the time follow-up was terminated for this clinical trial, several patients had not yet progressed or died. Their time to progression will remain unknown and not collected. | 4.5 [1 to NA] — At the time follow-up was terminated for this clinical trial, several patients had not yet progressed or died. Their time to progression will remain unknown and not collected.

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all eligible patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented.
Time Frame: Up to 3 years
Population: Participants with Complete or Partial response, were analyzed
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 (Prior Chemotherapy, PT) | Cohort 2 (Chemotherapy Naive, CN)
Number analyzed (Participants) | 3 | 10
months | 3.5 [3.2 to 11.6] | 12.1 [4.0 to 30.6]

5. Secondary Outcome: Number of Treatment Cycles Administered
Description: Number of treatment cycles administered is defined to be the number of treatment cycles administered until the patient is removed from treatment due to progression, toxicity, or refusal. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: cycles
Arm/Group | Cohort 1 (Prior Chemotherapy, PT) | Cohort 2 (Chemotherapy Naive, CN)
Number analyzed (Participants) | 34 | 39
cycles | 4 [1 to 10] | 4 [1 to 26]

ADVERSE EVENTS:
Time Frame: Adverse events are assessed during the Active Monitoring Phase prior to each cycle of treatment, during observation every 2 months until progression, and at time of progression; up to 2 years post-registration.
Description: This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) v3.0 for adverse event monitoring and reporting. All graded adverse events are reported.
Groups:
- Cohort 1 (Prior Chemotherapy, PT): chemotherapy for their metastatic disease receive 100 mg/m^2 paclitaxel albumin-stabilized nanoparticle formulation (ABI-007) IV over 30 minutes followed by AUC 2 carboplatin IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for at least 8 courses in the absence of disease progression or unacceptable toxicity.
- Cohort 2 (Chemotherapy Naive, CN): prior chemotherapy for their metastatic disease, patients receive 100 mg/m^2 paclitaxel albumin-stabilized nanoparticle formulation (ABI-007) IV over 30 minutes followed by AUC 2 carboplatin IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for at least 8 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Cohort 1 (Prior Chemotherapy, PT) | Cohort 2 (Chemotherapy Naive, CN)
Serious Adverse Events (participants affected / at risk) | 3/34 | 5/39
Other Adverse Events (participants affected / at risk) | 34/34 | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Prior Chemotherapy, PT) (N=34) | Cohort 2 (Chemotherapy Naive, CN) (N=39)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Prior Chemotherapy, PT) (N=34) | Cohort 2 (Chemotherapy Naive, CN) (N=39)
Hemoglobin decreased (Blood and lymphatic system disorders) | 29 (103) | 35 (139)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (8)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (3)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 22 (50) | 22 (48)
Vomiting (Gastrointestinal disorders) | 10 (12) | 10 (17)
Chest pain (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 30 (87) | 35 (154)
Fever (General disorders) | 3 (4) | 3 (5)
Localized edema (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (4) | 4 (5)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 9 (23) | 9 (13)
Lymphocyte count decreased (Investigations) | 2 (4) | 4 (8)
Neutrophil count decreased (Investigations) | 21 (70) | 28 (91)
Platelet count decreased (Investigations) | 18 (37) | 20 (46)
Weight loss (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 9 (18) | 10 (24)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (23) | 13 (30)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 20 (41) | 19 (76)
Taste alteration (Nervous system disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (7) | 8 (24)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes